CLINICAL TRIAL: NCT07089173
Title: The Effect-site Concentration of Remifentanil Blunting Endotracheal Intubation Responses During Anesthesia Induction With Lidocaine or Sufentanil Combined With Etomidate: A Randomized Controlled Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-112
Record Dates: First submitted 2025-07-08; First posted 2025-07-28 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-07

CONDITIONS: Hemodynamics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo group (Placebo Comparator)
  Interventions: Drug: Intravenous normal saline (NS 0.9)
- sufentanil group (Experimental)
  Interventions: Drug: intravenous sufentanil
- lidocaine group (Experimental)
  Interventions: Drug: Intravenous lidocaine

INTERVENTIONS:
Drug: Intravenous normal saline (NS 0.9) — Under target-controlled infusion (TCI) of remifentanil, anesthesia induction is performed using placebo (normal saline) combined with etomidate (0.3 mg/kg).
  Arms: placebo group
Drug: intravenous sufentanil — Under target-controlled infusion (TCI) of remifentanil, anesthesia induction is performed using sufentanil (0.2μg/kg) combined with etomidate (0.3 mg/kg).
  Arms: sufentanil group
Drug: Intravenous lidocaine — Under target-controlled infusion (TCI) of remifentanil, anesthesia induction is performed using lidocaine (1.5 mg/kg) combined with etomidate (0.3 mg/kg).
  Arms: lidocaine group

SUMMARY:
The aim of this study was to compare the effect-site target concentration (including EC₅₀ and EC₉₀) of remifentanil required to suppress cardiovascular responses to tracheal intubation during anesthesia induction with etomidate combined with either lidocaine or sufentanil.

DETAILED DESCRIPTION:
This study is a single-center, randomized controlled trial utilizing a modified sequential method to determine the effect site target concentration of remifentanil, including the median effective concentration (EC₅₀) and the 90% effective concentration (EC₉₀). The study population consists of ASA class I-II patients undergoing general anesthesia with endotracheal intubation. Patients will be randomly assigned to one of three groups: placebo group, lidocaine group, and sufentanil group. Patients in each group will receive anesthesia induction with a combination of either saline, lidocaine, or sufentanil along with etomidate, followed by target-controlled infusion of remifentanil. The primary outcome measure is the median effective target concentration of remifentanil in the effect site (EC₅₀) for suppressing the intubation response. Secondary outcomes include the 90% effective target concentration of remifentanil (EC₉₀), changes in mean arterial pressure (MAP), heart rate (HR), and bispectral index (BIS) before and after intubation. Each group is expected to enroll 33 patients, totaling 99 patients across all three groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgery under general anesthesia with endotracheal intubation;
* Classified as ASA physical status I-II.

Exclusion Criteria:

* Age <18 years or >65 years;
* Body mass index (BMI) >30 kg/m² or <18.5 kg/m²;
* Diagnosis of hypertension or severe cardiovascular diseases (including myocardial infarction, heart failure, atrial fibrillation, atrioventricular block, moderate-to-severe valvular diseases) or respiratory diseases (including acute exacerbation of chronic obstructive pulmonary disease, acute respiratory distress syndrome, acute asthma attack, moderate-to-severe pulmonary hypertension, severe pneumonia);
* Diagnosis of obstructive sleep apnea syndrome or history of difficult intubation or preoperatively anticipated difficult airway;
* Renal, hepatic or hematologic diseases;
* High risk of aspiration or reflux;
* Current use of analgesics for chronic pain or β-blockers for cardiovascular diseases;
* Current use of psychotropic medications;
* Contraindications to remifentanil or sufentanil, including: known hypersensitivity to any component of these drugs or other fentanyl analogues, current use of monoamine oxidase inhibitors, myasthenia gravis or conditions predisposing to respiratory depression, bronchial asthma or related disorders;
* Contraindications to lidocaine, including: known allergy to local anesthetics, concurrent Adams-Stokes syndrome, Wolff-Parkinson-White syndrome, or severe cardiac conduction block.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
The 50% effective effect-site target concentration (EC₅₀) of remifentanil for suppressing patients' tracheal intubation response | Through study completion, an average of 1 year.

SECONDARY OUTCOMES:
The 90% effective effect-site target concentration (EC₉₀) of remifentanil for suppressing patients' tracheal intubation response | Through study completion, an average of 1 year.
complications | Operative day, Postoperative day 1, Postoperative day 5.
  including excessive hemodynamic fluctuations, hypoxemia, coughing during induction, etomidate-induced myoclonus, opioid-related chest wall rigidity, and postoperative nausea and vomiting (PONV).

CONTACTS AND LOCATIONS:
Overall Officials: Tao Luo, Principal Investigator — Peking University Shenzhen Hospitai
Locations (1):
- Peking University Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee IW, Schraag S. The Use of Intravenous Lidocaine in Perioperative Medicine: Anaesthetic, Analgesic and Immune-Modulatory Aspects. J Clin Med. 2022 Jun 20;11(12):3543. doi: 10.3390/jcm11123543. PMID 35743617
- [Background] Guignard B, Menigaux C, Dupont X, Fletcher D, Chauvin M. The effect of remifentanil on the bispectral index change and hemodynamic responses after orotracheal intubation. Anesth Analg. 2000 Jan;90(1):161-7. doi: 10.1097/00000539-200001000-00034. PMID 10624998
- [Background] Gelberg J, Jonmarker C, Stenqvist O, Werner O. Intravenous boluses of fentanyl, 1 mug kg(-)(1), and remifentanil, 0.5 mug kg(-)(1), give similar maximum ventilatory depression in awake volunteers. Br J Anaesth. 2012 Jun;108(6):1028-34. doi: 10.1093/bja/aes029. Epub 2012 Mar 22. PMID 22440314
- [Background] Baldo BA. Toxicities of opioid analgesics: respiratory depression, histamine release, hemodynamic changes, hypersensitivity, serotonin toxicity. Arch Toxicol. 2021 Aug;95(8):2627-2642. doi: 10.1007/s00204-021-03068-2. Epub 2021 May 11. PMID 33974096
- [Background] Trujillo C, Rudd D, Ogutcu H, Dong F, Wong D, Neeki M. Objective Characterization of Opiate-Induced Chest Wall Rigidity. Cureus. 2020 Jun 5;12(6):e8459. doi: 10.7759/cureus.8459. PMID 32566433
- [Background] Oron AP, Souter MJ, Flournoy N. Understanding Research Methods: Up-and-down Designs for Dose-finding. Anesthesiology. 2022 Aug 1;137(2):137-150. doi: 10.1097/ALN.0000000000004282. PMID 35819863
- [Background] Burlacu CL, McKeating K, McShane AJ. Remifentanil for the insertion and removal of long-term central venous access during monitored anesthesia care. J Clin Anesth. 2011 Jun;23(4):286-91. doi: 10.1016/j.jclinane.2010.12.007. PMID 21663812
- [Background] Perez JJ, Strunk JD, Preciado OM, DeFaccio RJ, Chang LC, Mallipeddi MK, Deal SB, Oryhan CL. Effect of an opioid-free anesthetic on postoperative opioid consumption after laparoscopic bariatric surgery: a prospective, single-blinded, randomized controlled trial. Reg Anesth Pain Med. 2025 Sep 4;50(9):699-705. doi: 10.1136/rapm-2024-105632. PMID 38839427
- [Background] Hao Z, Jiang Z, Li J, Luo T. The effect-site concentration of remifentanil blunting endotracheal intubation responses in elderly patients during anesthesia induction with etomidate: a dose-exploration study. BMC Anesthesiol. 2025 Feb 13;25(1):70. doi: 10.1186/s12871-024-02844-8. PMID 39948474
- [Background] Jiang Z, Xiao J, Wang X, Luo T. The effect-site concentration of remifentanil blunting endotracheal intubation responses during anesthesia induction with etomidate: a dose-finding study. BMC Anesthesiol. 2023 Jun 28;23(1):225. doi: 10.1186/s12871-023-02165-2. PMID 37380959
- [Background] Albertin A, Casati A, Federica L, Roberto V, Travaglini V, Bergonzi P, Torri G. The effect-site concentration of remifentanil blunting cardiovascular responses to tracheal intubation and skin incision during bispectral index-guided propofol anesthesia. Anesth Analg. 2005 Jul;101(1):125-30, table of contents. doi: 10.1213/01.ANE.0000153012.35120.FE. PMID 15976218
- [Background] Misganaw A, Sitote M, Jemal S, Melese E, Hune M, Seyoum F, Sema A, Bimrew D. Comparison of intravenous magnesium sulphate and lidocaine for attenuation of cardiovascular response to laryngoscopy and endotracheal intubation in elective surgical patients at Zewditu Memorial Hospital Addis Ababa, Ethiopia. PLoS One. 2021 Jun 1;16(6):e0252465. doi: 10.1371/journal.pone.0252465. eCollection 2021. PMID 34061894
- [Background] Dunn LK, Durieux ME. Perioperative Use of Intravenous Lidocaine. Anesthesiology. 2017 Apr;126(4):729-737. doi: 10.1097/ALN.0000000000001527. No abstract available. PMID 28114177
- [Background] Yeganeh N, Roshani B, Latifi H, Almasi A. Comparison of target-controlled infusion of sufentanil and remifentanil in blunting hemodynamic response to tracheal intubation. J Inj Violence Res. 2013 Jul;5(2):101-7. doi: 10.5249/jivr.v5i2.325. Epub 2013 Feb 15. PMID 23416718
- [Background] Habib AS, Parker JL, Maguire AM, Rowbotham DJ, Thompson JP. Effects of remifentanil and alfentanil on the cardiovascular responses to induction of anaesthesia and tracheal intubation in the elderly. Br J Anaesth. 2002 Mar;88(3):430-3. doi: 10.1093/bja/88.3.430. PMID 11990278
- [Background] Forman SA. Clinical and molecular pharmacology of etomidate. Anesthesiology. 2011 Mar;114(3):695-707. doi: 10.1097/ALN.0b013e3181ff72b5. PMID 21263301
- [Background] Yoo KY, Jeong CW, Park BY, Kim SJ, Jeong ST, Shin MH, Lee J. Effects of remifentanil on cardiovascular and bispectral index responses to endotracheal intubation in severe pre-eclamptic patients undergoing Caesarean delivery under general anaesthesia. Br J Anaesth. 2009 Jun;102(6):812-9. doi: 10.1093/bja/aep099. Epub 2009 May 8. PMID 19429669
- [Background] Thompson JP, Hall AP, Russell J, Cagney B, Rowbotham DJ. Effect of remifentanil on the haemodynamic response to orotracheal intubation. Br J Anaesth. 1998 Apr;80(4):467-9. doi: 10.1093/bja/80.4.467. PMID 9640152
- [Background] Safavi M, Honarmand A. Attenuation of cardiovascular responses to laryngoscopy and tracheal intubation--intravenous sufentanil vs pethidine. Middle East J Anaesthesiol. 2008 Oct;19(6):1349-59. PMID 18942248
- [Background] Kayhan Z, Aldemir D, Mutlu H, Ogus E. Which is responsible for the haemodynamic response due to laryngoscopy and endotracheal intubation? Catecholamines, vasopressin or angiotensin? Eur J Anaesthesiol. 2005 Oct;22(10):780-5. doi: 10.1017/s0265021505001298. PMID 16211744